CLINICAL TRIAL: NCT06423807
Title: Preoperative Ondansetron Lozenge for Prevention of Post-Spinal Shivering in Caesarean Section: A Randomized Controlled Trial
Brief Title: Preoperative Ondansetron Lozenge for Prevention of Post-Spinal Shivering in Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36264PR642/4/24
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Ondansetron Lozenge; Post-Spinal Shivering; Cesarean Section

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Ondansetron lozenge) (Experimental): Patients will receive ondansetron lozenge 4 mg (Ondalenz ©), 2 hours before surgery as a study group.
  Interventions: Drug: Ondansetron lozenge
- Group C (Control) (No Intervention): Patients will not receive ondansetron as a control group.

INTERVENTIONS:
Drug: Ondansetron lozenge — Patients will receive ondansetron lozenge 4 mg (Ondalenz ©), 2 hours before surgery.
  Arms: Group S (Ondansetron lozenge)

SUMMARY:
The aim of this study is to estimate the role of ondansetron lozenge on prevention of post-spinal shivering in cesarean section.

DETAILED DESCRIPTION:
Spinal anesthesia (SA) is preferred for cesarean section (CS) compared with general anesthesia(GA) because of several advantages, including prevention of the potential risk of GA-related neurotoxicity.

Post-spinal shivering (PSS) could be a provocative factor for postoperative pain and its appropriate treatment prevents non-thermoregulatory tremors. Shivering also causes aggravating postoperative pain by stretching of sutures.

Ondansetron is a selective antagonist for receptor 5-hydroxytryptamine 3 and is very effective in the prevention and treatment of shivering intra- and post-operation. Ondansetron can affect the body temperature and shivering in rats since the balance of nor-epinephrine and 5-hydroxytryptamine (5-HT) in the preoptic-anterior hypothalamus controls the temperature set point.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 40 years.
* American Society of Anesthesiology (ASA) physical status II.
* Parturient women undergoing CS under spinal anesthesia.

Exclusion Criteria:

* Parturient women with any contraindication or hypersensitivity to the study drugs.
* Any history of cardiovascular diseases, psychosis, hypertension, fetal distress, cord prolapse initial.
* Temperature more than 38°C or less than 36°C.
* Body Mass Index (BMI)> 40 kg/m2.
* Medical history of alcohol or drug abuse.
* Parkinson's disease or any extrapyramidal disease.
* Intraoperative blood transfusion.
* History of chemotherapy treatment.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Parturient women undergoing cesarean section under spinal anesthesia
Enrollment: 60 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Incidence of shivering | 24 hours postoperatively
  Shivering will be graded during the intraoperative and postoperative period using the scale validated by Crossley and Mahajan and Tsai and Chu.
  0=No shivering, 1=Piloerection or peripheral vasoconstriction but no visible shivering, 2=Muscular activity in only one muscle group, 3=Muscular activity in more than one muscle group but not generalized shivering, 4=Shivering involving the whole body.
  Grades 3, and 4 shivering for at least 3 min will be considered positive, and maximum shivering will be considered if generalized shivering interfering with ECG monitoring or ability of the mother to hold the baby.

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV) | 24 hours postoperatively
  The incidence of nausea and vomiting will be evaluated through the Bellville scoring scale (lack of nausea and vomiting=0, nausea=1, nausea with belching=2, and vomiting=3).
Patients' satisfaction | 24 hours postoperatively
  • Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Adverse effects | 24 hours postoperatively
  Adverse events such as bradycardia, hypotension, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Elsharkawy, MD, Principal Investigator — Faculty of Medicine Tanta University, Egypt
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.